CLINICAL TRIAL: NCT06430021
Title: Study of the Value of HPG80 (circulating Progastrin) for the Diagnosis of Neuroendocrine Tumours in Patients with an NEM1 Mutation: the Progastrin-NEM1 Study
Brief Title: Study of the Value of HPG80 (circulating Progastrin) for the Diagnosis of Neuroendocrine Tumours in Patients with an MEN1 Mutation
Acronym: PRO-NEM1
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GOUDET BIODENA 2023
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Neuroendocrine Tumors; MEN1 Mutation
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patient: patients with proven MEN1, symptomatic or not
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — 8 mL blood sample in EDTA tube

SUMMARY:
Multiple Endocrine Neoplasia type 1 (MEN1) is an autosomal dominant disease with a high degree of penetrance (>80% of patients). It is caused by the presence of the MEN1 mutation located on chromosome 11q13. The prevalence of this mutation is estimated at approximately 1/30,000. This hereditary syndrome is characterized by the presence of tumours of the endocrine system (adenoma of the parathyroid, pituitary and adrenal glands, neuroendocrine tumors - NETs - of the endocrine pancreas, duodenum, lung or thymus), which threaten the health of these patients. Other malignant tumors such as breast cancer are also more common in patients with MEN1.

The clinical manifestations of MEN1 are linked to the location of the adenomas and NETs and their secretory products. Indeed, most NETs produce and secrete numerous peptide hormones (in the case of Insulinomas, Gastrinomas, VIPomas, Glucagonomas or PPomas for example). This causes a specific clinical syndrome, which can be detected in the blood serum. However, most NETs are "non-functional" tumors, which do not have specific secretions.

Among general tumor markers, chromogranin A (CgA) is widely used as a biomarker for monitoring NETs. CgA is a secretory protein released into the blood by neuroendocrine cells. However, the performance of CgA as a diagnostic biomarker is too limited to be used for the early identification of NETs, particularly in patients with MEN1.

This is why patients with MEN1 undergo regular biological and morphological examinations, at least once a year, to screen for the development of adenomas and NETs. However, CgA or hormone secretions assays, and imaging examinations (MRI, CT scan, or duodenopancratic endoscopic ultrasound (EUS)) are tedious and stressful for patients; in addition, they all have their limitations (poor performance for biological tests; irradiation for CT scan; need for anesthesia for endoscopic ultrasound, etc.). Consequently, there is a need for new markers to identify NETs in this population as early as possible.

Progastrin is a pro-hormone that, under physiological conditions, is matured into gastrin in the G cells of the antrum of the stomach. The role of gastrin is to stimulate gastric acid secretion during digestion. It also plays an important role in regulating cell growth in the gastric mucosa. In pathological situations, it has been shown that the GAST gene, which codes for progastrin, is over-expressed in human tumor cells of different origins, leading to the accumulation of progastrin within them. Tumor cells that are unable to mature progastrin into gastrin, either because the maturation enzymes are not expressed or are inhibited, will secrete it. This circulating progastrin is then called hPG80 (to differentiate it from intracellular progastrin) and is detectable in patient blood. hPG80 is a new biomarker for the detection of different types of cancer. It appears to be elevated in the early stages of the disease, potentially more so than other biomarkers such as circulating tumor DNA (ctDNA) or NETest. In addition, hPG80 is easily measured in plasma using the DxPG80.Lab ELISA (Progastrin Manufacturing). The analytical characteristics of this CE-marked in vitro diagnostic test have been published in the Analytical Methods journal. It has been validated in numerous studies of various cancers, including NET patients. In addition, a study conducted by the team at Progastrin Manufacturing (formerly ECS-Progastrin) showed that hPG80 was unequivocally present in the peripheral blood of patients with 11 different types of cancer, with a concentration significantly higher than that found in blood donors considered to be healthy. We therefore hypothesize that hPG80 could also be a biomarker for NETs in MEN1.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven MEN1, symptomatic or not, confirmed on the basis of the following international criteria (Thakker et al.):
* patients with an MEN1 mutation;
* patients belonging to an identified MEN1 family in which at least one first-degree relative has been affected and has at least one MEN1-related lesion;
* patients without a positive genetic test or a family history of the disease, but with at least two of the three main MEN1 lesions (parathyroid adenomas, duodenopancreatic NETs and pituitary tumours).
* Majors patients,
* Patients who have undergone thoracoabdominal imaging (MRI, and/or CT and/or somatostatin receptor imaging (PET or octreotide scan)) within 3 months prior to inclusion or are due to undergo imaging within 3 months of inclusion to document the presence of NETs,
* Regardless of the treatment they are receiving (treatment naïve or treated patient),
* Regardless of the type of disease associated with MEN1 (presence or absence of NET, adenoma....),
* Patients who did not object to taking part in the study.

Exclusion Criteria:

* Person not affiliated to national health insurance
* Person subject to a measure legal protection (curatorship, guardianship, family empowerment) or a court order
* Pregnant, parturient or breastfeeding mothers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be seen for follow-up consultations
Sampling Method: Non-Probability Sample
Enrollment: 297 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Presence of at least one significant NET vs. absence of significant NET or resected NET without relapse confirmed by thoracic-abdominal imaging | Within 3 months before or after inclusion.
  Significant NET = metastatic or progressive morphologically or supracentimetric NET of the pancreas, duodenum, lung/bronchus or thymus absence of significant NET = patient with sub-centimetric, stable and asymptomatic NET / with or without adenoma

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No